CLINICAL TRIAL: NCT03274310
Title: FluSAFE: Flu SMS Alerts to Freeze Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Melissa Stockwell, Associate Professor of Pediatrics and Population and Family Health, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAR0955; 1R01AI127812-01 (NIH)
Record Dates: First submitted 2017-09-04; First posted 2017-09-06 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Influenza; Acute Respiratory Infection; Influenza-like Illness
Keywords: Influenza; Text message; Influenza-like Illness; Acute Respiratory Infection
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surveillance + Education arm (Experimental): Receipt of educational text message about ways to decrease household transmission of influenza and other respiratory infections in addition to surveillance messages
  Interventions: Behavioral: Educational text messages
- Surveillance-only arm (No Intervention): No intervention solely surveillance messages

INTERVENTIONS:
Behavioral: Educational text messages — Educational text message about ways to decrease household transmission of influenza and other respiratory infections
  Arms: Surveillance + Education arm

SUMMARY:
Influenza infection results in an estimated 31 million outpatient visits, 55,000 to 974,200 hospitalizations, and 3,000 to 49,000 deaths. Membership in household in which someone else has influenza is the major risk factor for contracting influenza. The household secondary attack rate (SAR) is as high as 19% based on laboratory-confirmed influenza and 30% based on symptoms. Non-pharmaceutical preventive measures, including education, may play a role in decreasing transmission, but are only effective if started within 36 hours of symptom onset in index cases. Yet, most interventions are delayed because they are not initiated until care is sought. The investigators have demonstrated in one primarily Latino, urban community sample, that text messaging can be used to rapidly identify community members with influenza-like illness (ILI) early in an illness. This early identification would enable implementation of an educational intervention in the optimal time frame to reduce influenza transmission. Providing education within a text message is a proven successful strategy to influence behavior. Text messaging itself is scalable, low-cost, and can be used in low literacy populations. However, using text-message based surveillance to trigger a real-time text-message behavioral educational intervention to decrease household influenza transmission has not been assessed.

DETAILED DESCRIPTION:
The study will enroll approximately 400 households with ≥1 child recruited from four contiguous communities in New York City. Households will be randomized, stratified by community 1:1 to receive surveillance-only (no text message education) vs. surveillance plus text message educational intervention. For symptom surveillance, households in both arms will receive text messages 3x/week during each influenza season and report if someone in the household has ILI symptoms. For those in the educational intervention arm, when an ILI/acute respiratory infections (ARI) is reported, a series of educational text messages will be sent with information to decrease household transmission.

ELIGIBILITY:
Inclusion Criteria:

* ≥3 persons per household
* At least one person who is less than 18 years old
* English or Spanish speaking
* Household reporter has cell phone with text messaging capabilities
* Household reporter willing to use text messages to report
* Reside within study neighborhoods in New York City

Exclusion Criteria

* Intention to move away from New York City area in <12 months
* Language other than English or Spanish

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1918 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Stockwell, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: households
Period: Overall Study
Arm/Group | Surveillance + Education Arm | Surveillance-only Arm
Started | 959; 203 households | 959; 208 households
Completed | 959; 203 households | 959; 208 households
Not Completed | 0; 0 households | 0; 0 households

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Surveillance + Education Arm | Surveillance-only Arm | Total
Number analyzed (Participants) | 959 | 959 | 1918
Age, Customized [Count of Participants; unit: Participants]
  Age: <18 years | 468 | 448 | 916
  Age: 18 years and over | 491 | 511 | 1002
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 546 | 518 | 1064
  Male | 413 | 441 | 854
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 133 | 132 | 265
  Not Hispanic or Latino | 824 | 827 | 1651
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Laboratory-confirmed Influenza Infections
Description: One self-swab of the index case and self-swabs of other household members will be analyzed using reverse transcription polymerase chain reaction (RT-PCR) to identify household transmission of laboratory-confirmed influenza.
Time Frame: Up to 5 days
Measure: Mean (Standard Error); unit: infections
Arm/Group | Surveillance + Education Arm | Surveillance-only Arm
Number analyzed (Participants) | 959 | 959
infections | .22 (0.04) | .14 (0.05)

2. Secondary Outcome: Number of Cases of Household Members Meeting Symptomatic Criteria for ILI/ARI
Description: The CDC-provided case definition for ARI is presence of at least two of the following: 1) rhinorrhea/nasal congestion; 2) sore throat; 3) cough; 4) fever/feverishness; 5) myalgia. The ILI definition is at least two of the following signs and symptoms: fever, cough, headache, sore throat, or myalgia.
Time Frame: Up to 5 days
Measure: Mean (Standard Error); unit: infections
Arm/Group | Surveillance + Education Arm | Surveillance-only Arm
Number analyzed (Participants) | 959 | 959
infections | .20 (.01) | .19 (.01)

3. Secondary Outcome: Number of Infections of Non-influenza Respiratory Viruses
Description: This outcome will measure household transmission of non-influenza respiratory viruses. One self-swab of the index case and self-swabs of other household members will be analyzed using RT-PCR to identify household transmission of non-influenza respiratory viruses
Time Frame: Up to 5 days
Measure: Mean (Standard Error); unit: infections
Arm/Group | Surveillance + Education Arm | Surveillance-only Arm
Number analyzed (Participants) | 959 | 959
infections | .27 (.02) | .23 (.02)

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Surveillance + Education Arm | Surveillance-only Arm
All-Cause Mortality (participants affected / at risk) | 0/959 | 0/959
Serious Adverse Events (participants affected / at risk) | 0/959 | 0/959
Other Adverse Events (participants affected / at risk) | 0/959 | 0/959

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT03274310/Prot_SAP_000.pdf